CLINICAL TRIAL: NCT05663827
Title: Ruxolitinib Add-on in Steroid-refractory Graft-vs-host Disease After Allogeneic Stem Cell Transplantation: a Single Institutional Experience
Brief Title: Ruxolitinib as add-on Therapy in Steroid-refractory Graft-vs-host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yi-Lun Wang (Other)
Responsible Party: Sponsor-Investigator, Yi-Lun Wang, Principal investigator, Division of Hematology/Oncology, Department of Pediatrics, Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSR-1123
Record Dates: First submitted 2022-11-23; First posted 2022-12-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Steroid Refractory GVHD
Keywords: acute lymphoblastic leukemia; hematopoietic stem cell transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Cases with steroid-refractory GVHD would be given an add-on therapy of age/weight adjusted dosage of Ruxolitinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ruxolitinib add-on group (Experimental): Once diagnosed with steroid-refractory GVHD, after discussion with family, as per their willing, Ruxolitinib will be administered as add-on therapy. Its dose depends on participants' age and body weight. Usually a dosage of 5mg once per day will be applied as initiation and titrated in accordance with clinical response.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — A dosage of 5mg once daily will be applied as initiation. After one week use, dose escalation or de-escalation would depend on clinical response.
  Other Names: Jakavi

SUMMARY:
Steroid-refractory graft-vs-host disease (SR-GVHD) is a major cause of mortality after allogeneic hematopoietic stem cell transplantation (HSCT). We sought to evaluate the effect and safety of ruxolitinib (RUX) add-on in the treatment of patients with SR-GVHD.

DETAILED DESCRIPTION:
Nowadays, second-line treatment for SR-GVHD differs between centers and depends on the physician's experience. The agents commonly used as second and further lines of therapy include anti-thymocyte globulin, mycophenolate mofetil, calcineurin inhibitor, or extracorporeal photopheresis. However, the response varied. This study highlighted that corticosteroid (CS) is not a panacea for treating GVHD, and some patients with remission still experience further relapse. Additionally, the identification of multiple infections adds complexity.

Hope was supposed to come in 2019 after the Food and Drug Administration (FDA) approved RUX for the therapy of SR-GVHD in adult and pediatric patients > 12 years. RUX add-on should be withheld as the risks outweigh the benefits, especially for patients who developed scleroderma and bronchiolitis obliterans. RUX can be added on as needed for the treatment of GVHD, especially in patients receiving DLI as relapse therapy with the conversion from mixed chimerism to complete chimerism. Despite some studies showing the efficacy of RUX across affected organs, some other data bring the opposite results. Thus we conducted this study to reinforce the efficacy of RUX as an add-on therapy for SR-GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hematologic disorder

Exclusion Criteria:

* Those who are not applicable of receiving Ruxolitinib as immunodeficiency-modulation therapy
* Those who are actively encountering acute infectious illness

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
GI symptoms secondary to GVHD | 3 years
  Diarrhea event exceeds a frequency of 5 times a day
Skin symptoms secondary to GVHD | 3 years
  Skin rash extends more than 25% of body surface area

SECONDARY OUTCOMES:
Overall survival | 3 years
  From diagnosis of SR-GVHD to mortality due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Tang-Her Jaing, Study Director — Division of Hematology/Oncology, Department of Pediatrics, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Participants' basic information could be shared. Yet detailed one including morbidity or clinical course may not be exposed.

REFERENCES:
- [Result] Malard F, Huang XJ, Sim JPY. Treatment and unmet needs in steroid-refractory acute graft-versus-host disease. Leukemia. 2020 May;34(5):1229-1240. doi: 10.1038/s41375-020-0804-2. Epub 2020 Apr 3. PMID 32242050
- [Result] Wolff D, Fatobene G, Rocha V, Kroger N, Flowers ME. Steroid-refractory chronic graft-versus-host disease: treatment options and patient management. Bone Marrow Transplant. 2021 Sep;56(9):2079-2087. doi: 10.1038/s41409-021-01389-5. Epub 2021 Jul 3. PMID 34218265
- [Result] Przepiorka D, Luo L, Subramaniam S, Qiu J, Gudi R, Cunningham LC, Nie L, Leong R, Ma L, Sheth C, Deisseroth A, Goldberg KB, Blumenthal GM, Pazdur R. FDA Approval Summary: Ruxolitinib for Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease. Oncologist. 2020 Feb;25(2):e328-e334. doi: 10.1634/theoncologist.2019-0627. Epub 2019 Oct 22. PMID 32043777